CLINICAL TRIAL: NCT00109850
Title: Cetuximab Plus Cisplatin, Irinotecan and Thoracic Radiotherapy (TRT) for Locally Advanced (Non-Metastatic), Clinically Unresectable Esophageal Cancer: A Phase II Trial With Molecular Correlates
Brief Title: S0414 Cetuximab, Combo Chemo, and RT in Locally Advanced Esophageal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000426442; S0414 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Cisplatin; Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Cetuximab+Cisplatin+Irinotecan followed by radiation therapy (RT) in Cycle 3.
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: irinotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab — 400mg/m^2 loading dose, intravenous (IV) over 120 min, day 1 of cycle 1 only. 250mg/m^2 maintenance dose, IV over 60 min, Days 8 & 15 of Cycle 1 and Days 1, 8, and 15 of subsequent cycles.
  Other Names: Erbitux
Drug: cisplatin — 30mg/m^2, bolus intravenous (IV), on Days 1 & 8 of each cycle.
  Other Names: Platinol
Drug: irinotecan hydrochloride — 65mg/m^2, intravenous (IV) over 30 min, on Days 1 & 8 of each cycle.
  Other Names: CPT-11
Radiation: radiation therapy — The total dose to the prescription point will be 5,040 cGy given in 28 fractions. The patient will be treated with one fraction per day with all fields treated per day. 180 cGy will be delivered to the isocenter. The dose variation in the planning target volume (PTV) will be +7% and -5% of the prescription point dose.
  Other Names: RT; TRT

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of esophageal cancer by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cetuximab together with combination chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with combination chemotherapy and radiation therapy works in treating patients with locally advanced esophageal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year overall survival of patients with previously untreated, clinically unresectable, locally advanced squamous cell carcinoma or adenocarcinoma of the esophagus treated with cetuximab, cisplatin, irinotecan, and thoracic radiotherapy.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Determine the probability of objective response (confirmed and unconfirmed, complete and partial) in patients with measurable disease treated with this regimen.
* Determine the time to progression in patients with measurable disease treated with this regimen.
* Correlate, preliminarily, gene expression (RNA) levels and germline polymorphisms of genes involved in DNA repair (e.g., ECRCC-1 and XRCC-1), drug metabolism (e.g., UGT1A1), and the epidermal growth factor receptor (EGFR) pathway (e.g., EGFR, interleukin-8, and vascular endothelial growth factor) with response, time to progression, overall survival, and toxicity in patients treated with this regimen. (This will not be completed as this study was closed due to poor accrual.)

OUTLINE: This is a multicenter study.

Patients receive cetuximab intravenous (IV) over 1-2 hours on days 1, 8, and 15. Patients also receive cisplatin IV and irinotecan IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of course 3, patients undergo thoracic radiotherapy once daily 5 days a week for 5-6 weeks (total of 28 treatments).

After completion of study treatment, patients are followed at 4 weeks and then every 3-6 months for up to 5 years after study entry.

PROJECTED ACCRUAL: A total of 75-100 patients (75 with adenocarcinoma and 25 with squamous cell carcinoma) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (≥ 20 cm from the incisors*) or the gastroesophageal junction (confined to ≤ 2 cm into the gastric cardia)

  * Disease confined to the esophagus or peri-esophageal soft tissue
  * T4, M0 disease
  * Surgically unresectable disease by esophageal endoscopic ultrasonography OR medically unresectable disease

NOTE: *Patients with primary disease < 26 cm from the incisors must undergo bronchoscopy AND have negative cytology within the past 4 weeks

* Measurable or non-measurable disease by x-ray, CT scan and/or MRI, or physical examination within the past 4 weeks (for measurable disease) or within the past 6 weeks (for non-measurable disease)
* Tumor specimens available
* No recurrent disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* White Blood Cell (WBC) count ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL

Hepatic

* Albumin normal
* Bilirubin normal
* Alkaline phosphatase normal
* Serum glutamic oxaloacetic transaminase (SGOT) or Serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 times upper limit of normal

Renal

* Creatinine clearance > 50 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior severe reaction to monoclonal antibodies
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for esophageal cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for esophageal cancer
* No concurrent intensity modulated radiotherapy
* No concurrent cobalt-60

Surgery

* No prior surgical resection or attempted surgical resection of esophageal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R. Thomas, MD, Study Chair — OHSU Knight Cancer Institute; Charles D. Blanke, MD, FACP, Study Chair — OHSU Knight Cancer Institute; James L. Abbruzzese, MD, Study Chair — M.D. Anderson Cancer Center; Lisa Hammond, MD, Study Chair — The University of Texas Health Science Center at San Antonio; Vivek Mehta, MD, Study Chair — Swedish Cancer Institute at Swedish Medical Center - First Hill Campus
Locations (132):
- United States (132):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - Eden Medical Center, Castro Valley, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Saint Rose Hospital, Hayward, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Care Medical Center, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - CCOP - Santa Rosa Memorial Hospital, Sana Rosa, California
  - Sutter Solano Medical Center, Vallejo, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Watson Clinic, LLC, Lakeland, Florida
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 22
Eligible | 21
Eligible and Began Protocol Therapy | 21
Completed | 18
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 61.4 [43.0 to 83.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 2 Years
Description: Measured from time of registration to date of death due to any cause, or last contact date
Time Frame: 0-2 years
Population: All eligible patients who started treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cetuximab+Cisplatin+Irinotecan Followed by Radiation Therapy: Patients received four 21-day cycles of cetuximab 400 mg/m^2 (day 1, cycle 1), cetuximab 250 mg/m^2 (day 8, 15, cycle 1, then days 1, 8 and 15 for subsequent cycles), cisplatin 30 mg/m^2 (days 1 and 8, all cycles), and irinotecan 65 mg/m^2 (days 1 and 8, all cycles). Thoracic Radiotherapy (TRT) was administered at 1.8 Gy in 28 daily fractions to a total dose of 50.4 Gy, beginning on day 1 of cycle 3.
Arm/Group | Cetuximab+Cisplatin+Irinotecan Followed by Radiation Therapy
Number analyzed (Participants) | 21
percentage of participants | 33.3 [14.6 to 57.0]

2. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events after every two cycles of chemotherapy.
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Cetuximab+Cisplatin+Irinotecan Followed by Radiation Therapy
Number analyzed (Participants) | 21
Participants
  Albumin, serum-low (hypoalbuminemia) | 1
  Anorexia | 4
  CNS cerebrovascular ischemia | 1
  Calcium, serum-low (hypocalcemia) | 1
  Creatinine | 1
  Death not associated w/CTCAE term - Sudden death | 1
  Dehydration | 4
  Dermatology/Skin-Other (Specify) | 1
  Diarrhea | 5
  Dysphagia (difficulty swallowing) | 3
  Esophagitis | 2
  Fatigue (asthenia, lethargy, malaise) | 5
  Febrile neutropenia | 1
  Glucose, serum-high (hyperglycemia) | 1
  Hemoglobin | 3
  Leukocytes (total WBC) | 9
  Lymphopenia | 4
  Magnesium, serum-low (hypomagnesemia) | 1
  Nausea | 4
  Necrosis, GI - Colon/cecum/appendix | 1
  Neuropathy: sensory | 1
  Neutrophils/granulocytes (ANC/AGC) | 6
  Pain - Abdomen NOS | 1
  Pain - Esophagus | 1
  Perforation, GI - Colon | 1
  Potassium, serum-low (hypokalemia) | 2
  Rash: acne/acneiform | 1
  Renal failure | 1
  Sodium, serum-low (hyponatremia) | 1
  Thrombosis/thrombus/embolism | 1
  Typhlitis (cecal inflammation) | 1
  Vomiting | 3
  Weight loss | 1

3. Secondary Outcome: Objective Response (Confirmed and Unconfined, Complete and Partial)
Description: Complete response (CR) is complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. Normalization of markers and other abnormal lab values. Partial response (PR) applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. Confirmation of CR or PR means a repeat scan at least 4 weeks apart documented before progression or symptomatic deterioration.
Time Frame: at week 16, then every 3 months until progression
Population: All eligible patients who started treatment and were evaluable for response were included in assessing response estimates.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab+Cisplatin+Irinotecan Followed by Radiation Therapy
Number analyzed (Participants) | 17
percentage of participants | 17.6 [3.8 to 43.4]

4. Secondary Outcome: Progression Free Survival
Description: Measured from date of registration to date of first observation of progression or symptomatic deterioration. Patients last known to be alive and progression-free are censored at date of last contact.
Time Frame: 0 - 5 years
Population: All eligible patients who started treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab+Cisplatin+Irinotecan Followed by Radiation Therapy
Number analyzed (Participants) | 21
months | 6.4 [3.7 to 12]

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after every two cycles of chemotherapy.
Description: Only adverse events and serious adverse events that are possibly, probably or definitely related to study drug are reported.
Groups:
- Cetuximab+Cisplatin+Irinotecan Followed by RT in Cycle 3: Patients received four 21-day cycles of cetuximab 400 mg/m^2 (day 1, cycle 1), cetuximab 250 mg/m^2 (day 8, 15, cycle 1, then days 1, 8 and 15 for subsequent cycles), cisplatin 30 mg/m^2 (days 1 and 8, all cycles), and irinotecan 65 mg/m^2 (days 1 and 8, all cycles). Thoracic Radiotherapy (TRT) was administered at 1.8 Gy in 28 daily fractions to a total dose of 50.4 Gy, beginning on day 1 of cycle 3.
Arm/Group | Cetuximab+Cisplatin+Irinotecan Followed by RT in Cycle 3
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab+Cisplatin+Irinotecan Followed by RT in Cycle 3 (N=21)
Necrosis, GI - Colon/cecum/appendix (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Sudden death (General disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab+Cisplatin+Irinotecan Followed by RT in Cycle 3 (N=21)
Hemoglobin (Blood and lymphatic system disorders) | 10
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 15
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 8
Esophagitis (Gastrointestinal disorders) | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 19
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Pain - Esophagus (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 10
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
Rash: dermatitis associated with radiation - Chemoradiation (Injury, poisoning and procedural complications) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 2
Alkaline phosphatase (Investigations) | 4
Leukocytes (total WBC) (Investigations) | 14
Lymphopenia (Investigations) | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 14
Platelets (Investigations) | 8
Weight loss (Investigations) | 10
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 8
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 8
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 2
Taste alteration (dysgeusia) (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 13
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No